CLINICAL TRIAL: NCT00044265
Title: A Dose Escalation, Randomized, Double-blind Withdrawal Study of the Efficacy, Dose-response, and Safety of Ramipril for the Treatment of Hypertension in Children and Adolescents
Brief Title: Treatment of Pediatric Hypertension With Altace Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: K726-01-4002
Record Dates: First submitted 2002-08-23; First posted 2002-08-26 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: ACE inhibitor; high blood pressure; pediatric
MeSH Terms: conditions — Hypertension | interventions — Ramipril

INTERVENTIONS:
Drug: ramipril

SUMMARY:
Ramipril is an ACE inhibitor that has been marketed in the US for the treatment of hypertension since 1991. It has been shown to be effective in reducing both systolic and diastolic blood pressure in adults when used once daily. ACE inhibitors are frequently used to treat hypertension in children, however ramipril has not been extensively tested in children, and information regarding the efficacy and safety would therefore be of benefit to children. This study is designed to demonstrate the efficacy and safety of ramipril in the treatment of hypertension in children ages 6 through 16 years.

DETAILED DESCRIPTION:
In adults, common side effects include persistent dry mouth, dizziness, fatigue, and headache. Rare cases of angioedema have been reported. When used in pregnancy during the second and third trimesters, ACE inhibitors can cause injury and even death to the developing fetus. When pregnancy is detected, ramipril should be discontinued as soon as possible. Ramipril is contraindicated in patients who are hypersensitive to the product or have a history of angioedema related to previous treatment with an ACE inhibitor.

ELIGIBILITY:
Inclusion criteria:

* Males or females age 6 to 16 years. All female subjects ≥ 8 years of age must have a negative urine pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
* Weight ≥ 20 kg.
* Parents/guardians must be able to demonstrate their ability to use the home blood pressure device to monitor blood pressure.
* Sitting systolic blood pressure or sitting diastolic blood pressure ≥ the 95th percentile for age, gender and height; or diabetes mellitus or chronic renal insufficiency (as evidenced by GFR 40-70 mL/min/1.73 m2) and a sitting systolic blood pressure or sitting diastolic blood pressure ≥ the 90th percentile for age, gender, and height.

Exclusion criteria:

* Severe hypertension documented by (1) Sitting systolic blood pressure or sitting diastolic blood pressure more than 20 mmHg above the 95th percentile for age, gender, and height without antihypertensive therapy, (2) Sitting systolic blood pressure or sitting diastolic blood pressure more than 12 mmHg above the 95th percentile for age, gender, and height while receiving active therapy, or (3) hypertensive encephalopathy within the previous 5 months.
* Currently receiving more than one antihypertensive medication including: ACE inhibitors, angiotensin receptor inhibitors, beta blockers, calcium channel blockers, diuretics.
* Receiving lithium, potassium supplements, monoamine oxidase inhibitors, or major tranquilizers (Note: Stimulant medications for behavioral disorders, corticosteroids, and non-steroidal anti-inflammatory agents for chronic pain management are permitted during the trial provided the subject's dosage is anticipated to remain unchanged throughout the duration of the study.)
* A history of cardiomyopathy, clinically significant structural heart disease or atrioventricular conduction disturbance, sick sinus syndrome, atrial flutter, atrial fibrillation, clinically significant bradycardia or an accessory bypass tract, or clinical symptoms of congestive heart failure.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310
Dates: Start 2002-07; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sante Los Angeles, Los Angeles, California
  - Neufeld Medical Group, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Medical College of Georgia, Augusta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Nephrology and Hypertension Consultants, Park Ridge, Illinois
  - University of Louisville, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Univ of Missouri, Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - North Shore Univ Hospital c/o BRANY, Great Neck, New York
  - Montefiore Medical Center c/o BRANY, The Bronx, New York
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - PCTI at Columbus Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Le Bonheur Children's Hospital - Univ of Tennessee, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Medical Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin